CLINICAL TRIAL: NCT07375628
Title: Neurological and Cognitive Dysfunction Following CAR-T Treatment. ICANS and Beyond
Status: Not yet recruiting | Type: Observational
Sponsor: Karolinska University Hospital (Other)
Collaborators: Karolinska Institutet (Other); Kite, A Gilead Company (Industry)
Responsible Party: Principal Investigator, Ksenia Boriskina, Senior Consultant, Karolinska University Hospital
Other Study IDs: 2025-04301-01
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: CAR T Cell Therapy; ICANS; Cognitive and Executive Dysfunction
Keywords: Icans; CAR T cell therapy; Fatigue; Cognitive dysfunction; PET scan
MeSH Terms: conditions — Fatigue; Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood, saliva, bone marrow, cerobrospinal fluid
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Adult patients undergoing CAR T cell therapy in Region Stockholm: This project includes only adult patients (>20 years) in Region Stockholm. Participants will be patients with various hematologic diagnoses undergoing CAR-T. These patients are identified during routine care at ME CAST, Karolinska University Hospital.

SUMMARY:
This is a phase 4 non-interventional single center trial. We aim to prospectively include patients scheduled to undergo CAR-T therapy at ME CAST, Karolinska University Hospital Huddinge, to study ICANS. Because ICANS develops rapidly, inclusion during this potentially life-threatening phase would not be feasible; patients must therefore be enrolled before they start treatment. We aim to include patients who are clinically at high risk of developing ICANS. The risk of ICANS is assessed based on diagnosis, tumor burden, CAR-T product, and inflammatory status prior to treatment initiation. We plan to compare patients who develop ICANS grade 2-4 with patients who develop no ICANS or at most grade 1. Patients will undergo Positron Emission Tomography (PET) with two different tracers: (1) PBR28 for TSPO, which provides a measure of brain inflammation-this ligand binds to microglial cells-and (2) 11C-UCB-J for SV2A, which provides a measure of synaptic density in the brain. The results will be compared with magnetic resonance imaging. We will collect blood, bone marrow and cerebrospinal fluid (CSF) samples from this patient cohort. Samples will be taken from all patients before, during, and after CAR-T treatment. Participation in the study also includes computer-based cognitive testing, neuropsychological evaluation and genetic testing to determine whether the patient has receptors allowing binding of the TSPO radioligand used during PET imaging.

DETAILED DESCRIPTION:
Neurological symptoms after immune effector cell therapy are poorly understood, even though acute neurological adverse events have been reported for all CAR T-cell products. Adverse events affecting the central nervous system (CNS) during CAR-T-cell treatment-known as Immune Effector Cell-Associated Neurotoxicity Syndrome (ICANS)-typically occur about 4-10 days after treatment and cause symptoms such as confusion and speech difficulties. The incidence of ICANS ranges from as low as 2% to as high as 60%-70%. Despite many research projects and clinical trials, the pathogenesis of acute neurological toxicity remains unclear. Although the acute symptoms of ICANS are well characterized, little is known about long-term effects regarding fatigue and cognitive function after this treatment.

We aim to prospectively include patients scheduled to undergo CAR-T therapy at ME CAST, Karolinska University Hospital Huddinge, to study ICANS. Because ICANS develops rapidly, inclusion during this potentially life-threatening phase would not be feasible; patients must therefore be enrolled before they start treatment. We aim to include patients who are clinically at high risk of developing ICANS. The risk of ICANS is assessed based on diagnosis, tumor burden, CAR-T product, and inflammatory status prior to treatment initiation. Although the life-threatening phase may resolve within a few days thanks to rapid diagnostics and optimized treatment, some patients develop more long-lasting symptoms. These patients may experience reduced quality of life and difficulty returning to work and daily routines. Unfortunately, it is currently difficult to quantify and grade these symptoms, which complicates, for example, sickness certification or rehabilitation. Moreover, knowledge is very limited regarding the pathophysiological factors underlying symptoms such as fatigue and cognitive difficulties, and treatment options are limited.

Based on our results in allogeneic stem cell-transplanted patients and prior research on ICANS, our hypothesis is that clinical tools can predict high risk for ICANS and that long-term symptoms are caused by persistent low-grade inflammation in the brain after the acute phase. We believe that patients have dysregulated microglial cells and injury to synaptic function in neurons. Previous research has shown that a reduced number of connections between nerve cells (synapses) causes mental fatigue and cognitive difficulties in several psychiatric and neurodegenerative disorders.

We now plan to compare patients who develop ICANS grade 2-4 with patients who develop no ICANS or at most grade 1. Patients will undergo Positron Emission Tomography (PET) with two different tracers: (1) PBR28 for TSPO, which provides a measure of brain inflammation-this ligand binds to microglial cells-and (2) 11C-UCB-J for SV2A, which provides a measure of synaptic density in the brain. The results will be compared with magnetic resonance imaging. Understanding the relationship between neuroinflammation and synapse loss and how this can lead to cognitive difficulties may ultimately lead to new treatment methods. We will collect blood and cerebrospinal fluid (CSF) samples from this patient cohort. Blood samples will be taken from all patients before, during, and after CAR-T treatment. In the event of ICANS, a lumbar puncture will be performed according to clinical routine and CSF will be collected for microbiological analyses, cell counts, biochemistry, flow cytometry, etc., with the addition of research samples. CAR-T cells will be quantified in blood and CSF. During the acute phase, patients with ICANS will undergo neuroimaging with CT and/or MRI. Much of the above already forms part of routine diagnostics, which we now wish to analyze prospectively. Participation in the study also includes computer-based cognitive testing and genetic testing to determine whether the patient has receptors allowing binding of the TSPO radioligand used during PET imaging.

We will also use SWECARNET, our national Swedish CAR-T cell network, to improve knowledge about ICANS and implement it into standard care. The primary aim is to perform in-depth descriptive analyses in patients with ICANS grades 2-4 and 0-1. The scientific objective is to investigate synaptic density, inflammation, and activation of glial cells.

ELIGIBILITY:
Inclusion Criteria:

* Age > 20

  * Planned to undergo CAR-T treatment
  * No known prior CNS diseases or head trauma
  * Prior CNS involvement of lymphoma or acute lymphoblastic leukemia is allowed, provided it is well-controlled and treated at inclusion
  * Capable of receiving tailored information about the research project and signing informed consent

Exclusion Criteria:

* • Age under 20 years

  * The patient has previously indicated they wish to refrain from research participation
  * Another concurrent neuroinflammatory or neurodegenerative disease, or malignant disease (other than the underlying condition) in the central nervous system

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants will be patients with various hematologic diagnoses undergoing CAR-T. These patients are identified during routine care at ME CAST, Karolinska University Hospital. Only adults (over 20 years) will be included.
Sampling Method: Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2028-05 (Estimated); Study Completion 2029-05 (Estimated)

PRIMARY OUTCOMES:
To perform in deep descriptive analysis of patients developing ICANS grade 2-4 compared to patients with no ICANS or ICANS grade 1. | 2028
  The primary aim is to perform in-depth descriptive analyses in patients with ICANS grades 2-4 and 0-1. The scientific objective is to investigate synaptic density, inflammation, and activation of glial cells, which according to our hypothesis are linked to fatigue and cognitive dysfunction after ICANS. Our hypothesis is that these symptoms are caused by immune activation in the brain, which can be detected, among other methods, by PET imaging. We further hypothesize that this inflammation leads to altered neuronal connectivity with synaptic involvement.

CONTACTS AND LOCATIONS:
Overall Officials: Stephan Mielke, professor, Principal Investigator — Karolinska

IPD SHARING:
Plan to Share IPD: Undecided
to be discussed

REFERENCES:
- [Background] 1. Kazzi C, Kuznetsova V, Siriratnam P, Griffith S, Wong S, Tam CS, Alpitsis R, Spencer A, O'Brien TJ, Malpas CB, Monif M. Cognition following chimeric antigen receptor T-cell therapy: A systematic review. J Autoimmun. 2023 Nov;140:103126. doi: 10.1016/j.jaut.2023.103126. Epub 2023 Oct 12. PMID: 37837807. 2. Gust J, Ponce R, Liles WC, Garden GA and Turtle CJ (2020) Cytokines in CAR T Cell-Associated Neurotoxicity. Front. Immunol. 11:577027. doi: 10.3389/fimmu.2020.577027 3. Morbelli, S., Gambella, M., Raiola, A. M., Ghiggi, C., Bauckneht, M., Di Raimondo, T., Lapucci, C., Sambuceti, G., Inglese, M., & Angelucci, E. Brain FDG-PET findings in chimeric antigen receptor T-cell therapy neurotoxicity for diffuse large B-cell lymphoma. Journal of Neuroimaging 2023 DOI: 10.1111/jon.13135 4. Vinnakota, J.M., Biavasco, F., Schwabenland, M. et al. Targeting TGFβ-activated kinase-1 activation in microglia reduces CAR T immune effector cell-associated neurotoxicity syndrome. Nat Cancer 5, 1227-1249 (2024). https://doi.org/10.1038/s43018-024-00764-7 5. Chauveau, F., Winkeler, A., Chalon, S. et al. PET imaging of neuroinflammation: any credible alternatives to TSPO yet?. Mol Psychiatry 30, 213-228 (2025). https://doi.org/10.1038/s41380-024-02656-9 6. Vardy J, Wong K, Yi QL, Park A, Maruff P, Wagner L, Tannock IF. Assessing cognitive function in cancer patients. Support Care Cancer. 2006 Nov;14(11):1111-8. doi: 10.1007/s00520-006-0037-6. Epub 2006 Mar 15. PMID: 16538498. 7. Meyer JH, et al. Neuroinflammation in psychiatric disorders: PET imaging and promising new targets. Lancet Psychiatry. 2020 Dec;7(12):1064-1074. doi: 10.1016/S2215-0366(20)30255-8. Epub 2020 Oct 21. PMID: 33098761; PMCID: PMC7893630. 8. Kreisl WC, et al. PET imaging of neuroinflammation in neurological disorders. Lancet Neurol. 2020 Nov;19(11):940-950. doi: 10.1016/S1474-4422(20)30346-X. PMID: 33098803; PMCID: PMC7912433. 9. Masdeu JC, Pascual B, Fujita M. Imaging Neuroinflammation in Neurodegenerative Disorders